CLINICAL TRIAL: NCT02390557
Title: Persons With Disabilities Generating Quality Metrics to Inform Integrated Care
Brief Title: Persons With Disabilities Generating Quality Metrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Lisa Iezzoni, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2014000899
Record Dates: First submitted 2015-02-24; First posted 2015-03-17 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-04

CONDITIONS: Physical Disability; Chronic Mental Disorder
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: control v Survey v YESHealth
Who Masked: Participant, Care Provider
Masking Description: Randomization was performed at the level of primary care practice. Providers and patients were unaware of assignment to study arms
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control - Standard Practice (No Intervention): Standard measures of quality at baseline. No intervention reports sent to providers
- Survey (Experimental): Persons with Disabilities Quality Survey.PDQS Survey Reports Intervention.reports sent to providers of OneCare enrollees
  Interventions: Other: Survey
- YESHealth (Experimental): Arm 3: YESHealth Reports and PDQS Survey Reports sent to providers of OneCare enrollees
  Interventions: Other: Survey; Other: YESHealth

INTERVENTIONS:
Other: Survey — PDQS survey reports only
  Arms: Survey; YESHealth
Other: YESHealth — Arm 3: YESHealth and PDQS survey reports to providers
  Arms: YESHealth

SUMMARY:
No standard way exists to measure the quality of medical care or independent living long-term services and supports provided to persons with disabilities. This project will: provide a broader picture of how consumers with disabilities define care and care quality; measure the value of using consumers' expertise in developing, collecting, and assessing quality measures; and use this information to assist One Care providers in improving care delivered to their enrollees

DETAILED DESCRIPTION:
The aims of the project are as follows:

1. To work with persons with significant physical disabilities and serious and persistent mental illness to develop two new approaches to assess quality of care:

   Approach #1: We will survey enrollees about their experiences in One Care and their thoughts about the care they receive. This survey will also ask One Care enrollees about how they manage their care and what self-direction means to them. The survey will be called the Persons with Disabilities Quality Survey (PDQ-S), and it will be available in English and Spanish versions.

   Approach #2: Enrollees in One Care will provide information about their perceptions of care quality to a trained team of persons with disabilities who will report the information to One Care care teams. The goal of the activity is to support quality improvement in One Care through hearing the consumer's voice. This is called YES Health - Your Experience: Speak up for better health care.
2. We want to test how providing consumer informed and consumer directed quality information to One Care providers affects One Care quality.
3. We want to improve the ability of One Care enrollees to manage their own health care and to recognize and report quality problems

ELIGIBILITY:
Inclusion Criteria:

* One Care enrollee
* Permanent physical disability and/or serious mental illness
* Seen at designated practice site
* English or Spanish speaking

Exclusion Criteria:

* Persons with an intellectual or a developmental disability

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 451 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa I Iezzoni, MD, MSc, Principal Investigator — Mongan Institute Health Policy Center, Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The unit of randomization is the practice. In each wave, we selected survey participants who were patients in those practices. For wave 2 we report the cases from Wave 1 who completed the Wave 2 survey.
Units Other Than Participants: provider practice
Groups:
- Control - Standard Practice: Standard measures of quality as scheduled through One Care demonstration
- Survey Arm: Consumer surveyed with Persons with Disabilities Quality Survey (PDQ-S) Results given to provider along with standard quality metric data as scheduled through One Care
- YES Health: Initiative created by persons with disabilities for persons with disabilities to actively engage in collecting, analyzing and reporting on quality of care from the consumer perspective. The purpose is to engage eligible enrollees to answer brief surveys surrounding various themes about the care and experiences they receive through One Care. Subsequent brief, actionable reports are fed back to primary care provider practices randomized to this arm.
  YES Health: Intervention Arm
Period: Wave 1
Arm/Group | Control - Standard Practice | Survey Arm | YES Health
Started | 160; 9 provider practice | 156; 9 provider practice | 135; 9 provider practice
Completed | 160; 9 provider practice | 156; 9 provider practice | 135; 9 provider practice
Not Completed | 0; 0 provider practice | 0; 0 provider practice | 0; 0 provider practice
Period: Wave 2
Arm/Group | Control - Standard Practice | Survey Arm | YES Health
Started | 160; 9 provider practice | 156; 9 provider practice | 135; 9 provider practice
Completed | 88; 9 provider practice | 115; 9 provider practice | 112; 9 provider practice
Not Completed | 72; 0 provider practice | 41; 0 provider practice | 23; 0 provider practice
Not completed — Survey non-respondent | 72 | 41 | 23

BASELINE CHARACTERISTICS:
Population: The baseline analysis population participants are the respondents to the Wave 1 survey who enrolled in the study by completing the baseline survey
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Standard Practice | Survey Arm | YES Health | Total
Number analyzed (Participants) | 160 | 156 | 135 | 451
Age, Categorical [Count of Participants; unit: Participants] — Population: Wave 2 data are for the participants who completed both Wave 1 and Wave 2 surveys
  Participants
    Wave 1: <=18 years | 0 | 0 | 0 | 0
    Wave 1: Between 18 and 65 years | 160 | 156 | 135 | 451
    Wave 1: >=65 years | 0 | 0 | 0 | 0
    Wave 2: number analyzed (Participants) | 88 | 115 | 112 | 315
    Wave 2: <=18 years | 0 | 0 | 0 | 0
    Wave 2: Between 18 and 65 years | 88 | 115 | 112 | 315
    Wave 2: >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Wave 1 row shows all participants who enrolled at baseline. The Wave 2 row shows all participants from wave 1 who completed the Wave 2 survey, thus providing data for the pre post comparisons in each study arm
  Participants
    Wave 1: Female | 92 | 83 | 73 | 248
    Wave 1: Male | 68 | 73 | 62 | 203
    Wave 2: number analyzed (Participants) | 88 | 115 | 112 | 315
    Wave 2: Female | 46 | 61 | 61 | 168
    Wave 2: Male | 42 | 54 | 51 | 147
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Wave 1 data are for enrolled subjects at Baseline Wave 2 data are for those who enrolled in Wave 1 who completed Wave 2 surveys for longitudinal pre post analyses
  Participants
    Wave 1: White | 87 | 63 | 53 | 203
    Wave 1: Black | 9 | 25 | 25 | 59
    Wave 1: Hispanics | 53 | 53 | 43 | 149
    Wave 1: Other | 11 | 15 | 14 | 40
    Wave 2: number analyzed (Participants) | 88 | 115 | 112 | 315
    Wave 2: White | 36 | 47 | 46 | 129
    Wave 2: Black | 14 | 18 | 18 | 50
    Wave 2: Hispanics | 30 | 39 | 38 | 107
    Wave 2: Other | 8 | 11 | 10 | 29
Disability Type [Count of Participants; unit: Participants] — Population: Wave 1 data are for baseline enrollees Wave 2 data are for Wave 1 enrollees who also completed Wave 2 survey
  Participants
    Wave 1: Significant Physical Disability | 60 | 64 | 51 | 175
    Wave 1: Severe Mental Illness | 100 | 92 | 84 | 276
    Wave 2: number analyzed (Participants) | 88 | 115 | 112 | 315
    Wave 2: Significant Physical Disability | 47 | 40 | 41 | 128
    Wave 2: Severe Mental Illness | 41 | 75 | 71 | 187

OUTCOME MEASURES:

1. Primary Outcome: Improved Quality of Care
Description: % who agree that their quality of care Is better, the same or worse than before
Time Frame: 12 months
Population: 315 participants completing wave 1 and wave 2 surveys
Measure: Count of Participants; unit: Participants
Groups:
- Control - Standard Practice: Control group with no intervention
Arm/Group | Control - Standard Practice | Survey Arm | YES Health
Number analyzed (Participants) | 88 | 115 | 112
Participants | 45 | 68 | 53
Statistical Analysis 1: Comparison: Control - Standard Practice vs Survey Arm; we had a prior hypothesis that the survey intervention would be associated with a larger increase in perceived quality of health care compared with control from Wave 1 to Wave 2; Test type: Superiority; p = 0.074, Chi-squared, Corrected; Mean Difference (Final Values) = 10.7
Statistical Analysis 2: Comparison: Control - Standard Practice vs YES Health; We compared change in perception of quality of health care between Control v YES Health, wave 1 v Wave 2; Test type: Superiority; p = .069, Chi-squared, Corrected; Mean Difference (Final Values) = 7.4

ADVERSE EVENTS:
Time Frame: 1 year
Description: We measured adverse events as reports of events from participants at time of survey or in the intervening period.
  These were surveys, no adverse events were reported by participants or next of kin
Arm/Group | Control - Standard Practice | Survey Arm | YES Health
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/156 | 0/135
Serious Adverse Events (participants affected / at risk) | 0/160 | 0/156 | 0/135
Other Adverse Events (participants affected / at risk) | 0/160 | 0/156 | 0/135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No